CLINICAL TRIAL: NCT06354049
Title: Reiki Therapy to Improve Key Symptoms in Integrative Oncology Clinic (REIKI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3Z24
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cancer Pain; Oncology Pain
Keywords: Reiki
MeSH Terms: conditions — Cancer Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reiki therapy (Experimental): This is a feasibility single arm trial of Reiki for oncology participants.
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Reiki — Reiki, originating in Japan, is a biofield therapy where a skilled practitioner places their hands on or above the body of the recipient or themselves to induce relaxation and promote healing.

SUMMARY:
The purpose of this research is to investigate the delivery of Reiki to integrative oncology patients and assess its potential for improving cancer-related symptoms in this population.

DETAILED DESCRIPTION:
Reiki is a biofield therapy originating in Japan, in which a trained practitioner places their hands on or above the body of a receiver or themselves to generate a relaxation and healing response. Systematic reviews and meta-analyses report Reiki to be effective for improving psychological and physical health symptoms. With respect to adults with cancer, Reiki has been shown to improve participants' relaxation, pain, fatigue, sleep, anxiety, stress, and wellbeing/quality of life compared to care as usual. However, one study showed no improvement in comfort and wellbeing in those receiving Reiki compared to sham Reiki control, but those receiving Reiki reported improvements above usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 89.
* Neoplasm diagnosis (i.e., ICD-10 C00 - D49) confirmed in electronic health record (EHR)/Caisis
* Receiving care at a UH Connor Whole Health Integrative Oncology Clinic.
* Reporting at least three ESAS symptoms ≥4/10 at baseline screening including fatigue and ≥2 other symptoms on the 9-item questionnaire.
* Able to speak and understand English.
* Has an email address, and access to a computer with internet and/or a mobile device with a functioning data plan

Exclusion Criteria:

* Significant cognitive impairment that has not been corrected.
* Significant visual impairment that has not been corrected.
* Unable to provide informed consent.
* Active psychosis.
* Pregnancy.
* Metastatic disease.
* Reiki therapy within 3 months of study enrollment
* Active immunotherapy, chemotherapy, or radiation treatment, or completed within 3 months before study start. Aromatase inhibitors and tamoxifen are exceptions.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Recruitment rate as measured by the percentage of participants enrolled | 8 weeks post enrollment
  Calculated by total number of participants enrolled/ total number of participants eligible and 90% is considered successful for the recruitment rate.
Retention rate as measured by the number of participants retained until the final survey point | 8 weeks post enrollment
  Calculated by number of participants retained until the final survey time point / number of participants enrolled. 70% of participant retention until the final survey time point will be considered successful.
Attendance rate as measured by number of sessions attended per 6 sessions | 8 weeks post enrollment
  Total number of sessions attended per 6 sessions. Attendance rate of >/= 70% will be considered successful
Protocol adherence rate as measured by the number of participants treated in manner consistent with the intervention | 8 weeks post enrollment
  Number of participants treated in manner consistent with intervention/total number of participants enrolled
Acceptability as measured by the patient mean of participant satisfaction survey | 8 weeks post enrollment
  As assessed by participants mean for the Participants' satisfaction survey with the Reiki sessions, measured on a scale from 0 (Not at all satisfied) to 10 (Completely satisfied)
Data completeness rate | 8 weeks post enrollment
  Data completeness of >/= 90% is considered satisfactory

SECONDARY OUTCOMES:
Patient-reported outcomes as measured by PROMIS-29(Patient-Reported Outcomes Measurement Information System) score | Baseline, 8 weeks
  Changes from baseline in Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Activities, Pain Interference all measured by T-score, a 11 point numerical rating scale, with higher scores representing more pain calculated from a 5 point Likert scale, with higher scores representing more of the concept being measured.
Patient-reported outcomes as measured by ESAS(Edmonton Symptom Assessment System) scale | Upto 8 weeks
  The rate of intensity of common cancer symptoms, including pain, nausea, anxiety, fatigue, and well-being as measured using ESAS scale of 0 to 10 where, 0 is no pain to 10 as worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Rao, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
When sharing IPD via open access, the lack of restrictions leads to greater risk of re-identifying individuals. Data could be inappropriately merged with other data to facilitate re-identification.The small study population makes this more likely. On the other hand, sharing IPD via controlled access is burdensome. It requires resources that the investigator does not have (setting up the infrastructure and policies, administering and reviewing data requests, preparing data and distributing data). The personnel time for such an endeavor was not budgeted nor does the investigator have the financial resources to include it in the study budget